CLINICAL TRIAL: NCT02993211
Title: Transurethral En Bloc Versus Standard Resection of Bladder Tumour: A Multi-centre Randomised Controlled Trial (EB-StaR Study).
Brief Title: Transurethral En Bloc Versus Standard Resection of Bladder Tumour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other); North District Hospital (Other); Our Lady of Maryknoll Hospital (Other); Pok Oi Hospital (Other); The University of Hong Kong (Other); Tseung Kwan O Hospital, Hong Kong (Other); Tuen Mun Hospital (Other Government); Tung Wah Hospital (Other); United Christian Hospital (Other); Princess Margaret Hospital, Hong Kong (Other Government); Caritas Medical Centre, Hong Kong (Other); Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Jeremy Yuen Chun TEOH, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRE Ref. No. 2016.553
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Transurethral resection; En bloc resection; TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard resection (Active Comparator): For patients undergoing bipolar transurethral standard resection, bladder tumour is resected in a piecemeal manner.
  Interventions: Device: Bipolar transurethral standard resection
- En bloc resection (Experimental): For patients undergoing bipolar transurethral en bloc resection, bladder tumour is resected and removed in one piece.
  Interventions: Device: Bipolar transurethral en bloc resection

INTERVENTIONS:
Device: Bipolar transurethral standard resection — Olympus TURis Bipolar HF-resection electrode (Model: WA22306D)
  Arms: Standard resection
Device: Bipolar transurethral en bloc resection — Olympus TURis Bipolar HF-resection electrode (Model: WA22306D)
  Arms: En bloc resection

SUMMARY:
Conventionally, transurethral standard resection (SR) of bladder tumour is performed in a piecemeal manner. Transurethral en bloc resection (EBR) has been described as an alternate surgical technique in bladder tumour resection. By preventing tumour fragmentation and ascertaining complete tumour resection by histological assessment of the EBR specimen, we hypothesized that EBR could reduce disease recurrence as compared to SR.

DETAILED DESCRIPTION:
Bladder cancer is the 9th most commonly diagnosed cancer in men worldwide, with a standardized incidence rate of 9.0 per 100,000 person-years for men and 2.2 per 100,000 person-years for women. In Hong Kong, more than 400 new cases of bladder cancer are diagnosed every year. It is a common and important disease which carries a significant burden to the health medical system.

For patients who are diagnosed to have bladder tumours upon flexible cystoscopy, transurethral resection of bladder tumour (TURBT) should be offered. Being a minimally invasive procedure, it has become the standard for the initial management of bladder cancer. This operation aims to ascertain the diagnosis, to correctly stage the tumour (T-stage) and to cure the disease in the case of non-muscle-invasive bladder cancer (NMIBC). However, in a combined analysis of 2,596 patents from 7 randomised controlled trials in patients with NMIBC, it was shown that 1-year recurrence rate ranged from 15-61%, and 5-year recurrence rate ranged from 31-78%. Despite possible complete tumour resection during TURBT, the oncological control of NMIBC is far from satisfactory.

There are two main problems with the conventional standard resection (SR) procedure. First, the bladder tumour is resected in a piecemeal manner. This results in tumour fragmentation and floating tumour cells inside the bladder. The tumour cells may re-implant on to the bladder wall and lead to early disease recurrence. Second, 'complete tumour resection' is often determined by endoscopic vision only. Due to the inherited nature of piecemeal resection, it is not possible to assess the resection margin by histological means. The charring effect to the resection bed may also hinder the judgement of a 'complete tumour resection'. Routine second-look TURBT has been advocated for selected patients (Any presence of T1 disease, G3 disease, or any absence of detrusor muscle in the first TURBT specimen) even after a 'complete tumour resection' during the first TURBT. Second-look TURBT has been shown to detect residual disease in 33-55% of the patients and upstaging of disease in 4-45% of the patients. These results highlighted the limitations of TURBT in ascertaining complete tumour resection.

Transurethral en bloc resection (EBR) has been described as an alternate surgical technique in bladder tumour resection. By preventing tumour fragmentation and ascertaining complete tumour resection by histological assessment of the EBR specimen, we hypothesized that EBR could reduce disease recurrence as compared to SR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old with informed consent

Exclusion Criteria:

* Bladder tumour base with maximal dimension of >3cm (Anticipated difficulty in retrieving the specimen en bloc)
* Bladder tumour detected during intravesical BCG therapy (BCG failure warrants more aggressive treatment, i.e. radical cystectomy)
* Histological diagnosis other than NMIBC
* Presence or prior history of upper urinary tract malignancy
* ECOG performance status ≥ 3 (Confined to bed or chair more than 50% of waking hours)
* ASA III or above (Patient with severe systemic disease)
* History of bleeding disorder or use of anti-coagulants
* Pregnancy
* Presence of other active malignancy
* Life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
One-year recurrence rate | One year after the allocated treatment
  Rate of disease recurrence one year after the operation

SECONDARY OUTCOMES:
Detrusor muscle sampling rate | One week after the allocated treatment
  Rate of presence of detrusor muscle in the pathological specimen
Occurrence of obturator reflex | Intra-operative
  Number of participants with obturator reflex encountered by the operating surgeon during the operation
Operative time | Immediately post-operative
  Duration of operation
Rate of mitomycin C instillation | One day after the allocated treatment
  Rate of mitomycin C instillation given after the operation
Hospital stay | Three days after the allocated treatment
  Patients undergoing transurethral resection surgery have an average hospital stay of three days.
30-day complications | Thirty days after the allocated treatment
  Complications which occur within 30 days after the operation
Residual disease upon second look transurethral resection surgery | Seven weeks after the allocated treatment
  Second look transurethral resection surgery is expected to perform within six weeks after the allocated treatment and one more week is allowed for histological assessment of the second look transurethral resection specimen. Residual disease is measured by the number of participants with the presence of urothelial carcinoma in the second look transurethral resection specimen.
Upstaging of disease upon second look transurethral resection surgery | Seven weeks after the allocated treatment
  Second look transurethral resection surgery is expected to perform within six weeks after the allocated treatment and one more week is allowed for histological assessment of the second look transurethral resection specimen. Upstaging of disease is measured by the number of participants with upstaging of disease from non-muscle-invasive bladder cancer to muscle-invasive bladder cancer in the second look transurethral resection specimen.
One-year progression rate | One year after the allocated treatment
  Rate of disease progression one year after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy YC Teoh, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (13):
- Hong Kong (13):
  - Caritas Medical Centre, Hong Kong
  - Kwong Wah Hospital, Hong Kong
  - North District Hospital, Hong Kong
  - Our Lady of Maryknoll Hospital, Hong Kong
  - Pok Oi Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tseung Kwan O Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Tung Wah Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208
- [Background] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Background] Grimm MO, Steinhoff C, Simon X, Spiegelhalder P, Ackermann R, Vogeli TA. Effect of routine repeat transurethral resection for superficial bladder cancer: a long-term observational study. J Urol. 2003 Aug;170(2 Pt 1):433-7. doi: 10.1097/01.ju.0000070437.14275.e0. PMID 12853793
- [Background] Divrik RT, Sahin AF, Yildirim U, Altok M, Zorlu F. Impact of routine second transurethral resection on the long-term outcome of patients with newly diagnosed pT1 urothelial carcinoma with respect to recurrence, progression rate, and disease-specific survival: a prospective randomised clinical trial. Eur Urol. 2010 Aug;58(2):185-90. doi: 10.1016/j.eururo.2010.03.007. Epub 2010 Mar 19. PMID 20303646
- [Background] Jahnson S, Wiklund F, Duchek M, Mestad O, Rintala E, Hellsten S, Malmstrom PU. Results of second-look resection after primary resection of T1 tumour of the urinary bladder. Scand J Urol Nephrol. 2005;39(3):206-10. doi: 10.1080/00365590510007793-1. PMID 16127800
- [Background] Lazica DA, Roth S, Brandt AS, Bottcher S, Mathers MJ, Ubrig B. Second transurethral resection after Ta high-grade bladder tumor: a 4.5-year period at a single university center. Urol Int. 2014;92(2):131-5. doi: 10.1159/000353089. Epub 2013 Aug 23. PMID 23988813
- [Background] Vasdev N, Dominguez-Escrig J, Paez E, Johnson MI, Durkan GC, Thorpe AC. The impact of early re-resection in patients with pT1 high-grade non-muscle invasive bladder cancer. Ecancermedicalscience. 2012;6:269. doi: 10.3332/ecancer.2012.269. Epub 2012 Sep 18. PMID 22988482
- [Background] Ukai R, Kawashita E, Ikeda H. A new technique for transurethral resection of superficial bladder tumor in 1 piece. J Urol. 2000 Mar;163(3):878-9. PMID 10687997
- [Background] Kramer MW, Rassweiler JJ, Klein J, Martov A, Baykov N, Lusuardi L, Janetschek G, Hurle R, Wolters M, Abbas M, von Klot CA, Leitenberger A, Riedl M, Nagele U, Merseburger AS, Kuczyk MA, Babjuk M, Herrmann TR. En bloc resection of urothelium carcinoma of the bladder (EBRUC): a European multicenter study to compare safety, efficacy, and outcome of laser and electrical en bloc transurethral resection of bladder tumor. World J Urol. 2015 Dec;33(12):1937-43. doi: 10.1007/s00345-015-1568-6. Epub 2015 Apr 25. PMID 25910478